CLINICAL TRIAL: NCT06928311
Title: Examining the Influence of Biophilic Design on College Students' Exercise Performance: A Crossover Study
Brief Title: This Study Explores Whether Adding Natural Elements Like Plants and Sunlight to Indoor Gyms Makes Exercise Feel Easier, More Enjoyable, and Improves Performance. By Comparing Workouts in Nature-inspired and Plain Gym Settings, it Aims to Find Better Ways to Design Fitness Spaces in Cities.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 6530
Record Dates: First submitted 2025-04-01; First posted 2025-04-15 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Biophilic Environmental Design; Traditional Exercise Design
Keywords: Exercise; Biophilia; Environmental Design; Mood; Exercise Enjoyment
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into the biophilia group or the traditional group - that will be the environment that they start in. They will then go through a week wash out and then will go into the other environment for their exercise test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biophilic Design (Experimental): The exercise environment will be designed with nature elements, real and artificial plants, a landscape wall paper, simulated sunlight, and nature sounds.
  Interventions: Other: Exercise Environment
- Traditional Exercise Environment (Experimental): The exercise environment will be designed like a traditional indoor gym setting. With a treadmill at the center and no other purposeful design elements.
  Interventions: Other: Exercise Environment

INTERVENTIONS:
Other: Exercise Environment — This intervention focused around the environmental design of the exercise room.

SUMMARY:
The goal of this observational study is to examine whether exercising in a biophilic environment - a space designed to include natural elements like real plants, simulated sunlight, nature sounds, and outdoor views - can improve exercise performance and enjoyment compared to a standard indoor gym environment in male college students age 18-25 who have regularly exercised prior.

The main question it aims to answer is: "Can biophilic design enhance the physical and mental benefits of indoor exercise?"

Researchers will compare the two environments to see if there is any changes in exercise performance and enjoyment for each participant.

Participants will complete a treadmill fitness test in both settings to compare physical outcomes like maximal aerobic capacity, so the maximal amount of oxygen one can use during exercise, as well as perceived effort. After each treadmill test participants will be given surveys where they will be asked to evaluate their mood and enjoyment in that environment.

ELIGIBILITY:
Inclusion Criteria:

* Men between 18 and 25 years

Exclusion Criteria:

* Resting BP greater than 140/90
* Resting HR greater than 100 bpm
* BMI greater than 30 kg/m^2
* inability to exercise at moderate to vigorous intensities
* major illness/health complication in the past

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2025-04-04 (Actual); Primary Completion 2025-10-16 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Maximal Aerobic Capacity (VO2Max) | Testing Day 1
  This will be taken using a K5 metabolic cart measuring breath by breath
Maximal Aerobic Capacity (VO2Max) | Testing Day 2
  This will be taken using a K5 metabolic cart measuring breath by breath
Rate of Perceived Exertion | Every minute during testing day 1
  Participants will rate their perceived exertion every minute during the test and recovery period on a 6-20 scale.
Rate of Perceived Exertion | Every minute during testing day 2
  Participants will rate their perceived exertion every minute during the test and recovery period on a 6-20 scale.
Mood and Enjoyment Survey | Post Test Day 1
  Participants will receive a paper survey on mood and enjoyment to complete.
Mood and Enjoyment Survey | Post Test Day 2
  Participants will receive a paper survey on mood and enjoyment to complete.
VO2 Plateau Duration | Post Test Day 1
  The time at which the participant is exercising at near maximal capacity.
VO2 Plateau Duration | Post Test Day 2
  The time at which the participant is exercising at near maximal capacity.

SECONDARY OUTCOMES:
Heart Rate | During Testing Day 1 and 2
  Taken using a Garmin HR chest strap.

CONTACTS AND LOCATIONS:
Overall Officials: Kaigang Li, Principal Investigator — Colorado State University
Locations (1):
- Colorado State University Cardio Room (Moby Arena 134), Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No